CLINICAL TRIAL: NCT01940146
Title: Efficacy and Safety of SPARC1310 in Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLR_13_10
Record Dates: First submitted 2013-09-06; First posted 2013-09-12 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SPARC Placebo (Placebo Comparator)
  Interventions: Drug: SPARC Placebo
- SPARC1310 I (Experimental)
  Interventions: Drug: SPARC1310 I
- SPARC1310 II (Experimental)
  Interventions: Drug: SPARC1310 II
- SPARC1310 III (Experimental)
  Interventions: Drug: SPARC1310 III

INTERVENTIONS:
Drug: SPARC Placebo — Placebo
  Arms: SPARC Placebo
Drug: SPARC1310 I — SPARC1310 I
  Arms: SPARC1310 I
Drug: SPARC1310 II — SPARC1310 II
  Arms: SPARC1310 II
Drug: SPARC1310 III — SPARC1310 III
  Arms: SPARC1310 III

SUMMARY:
The study will assess the efficacy and safety of SPARC1310 when compared to placebo and active control

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 65 years with history of seasonal allergic rhinitis
* Participants able to understand and willing to sign the informed consent form

Exclusion Criteria:

* Anotomical deviations of the nasal septum that significantly impair ventilation or airflow
* Pregnant or nursing women
* Positive serology for infectious disease (Hepatitis B or C, HIV) at screening
* Parallel participation in another current investigational study, participation in a study within less than 30 days prior to study entry, or previous participation in this same study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shravanti Bhowmik, MD, Study Director — Sun Pharma Advanced Research Company Limited
Locations (1):
- SPARC Site 1, Kingston, Canada

REFERENCES:
- [Derived] Ellis AK, Steacy LM, Joshi A, Bhowmik S, Raut A. Efficacy of the novel nasal steroid S0597 tested in an environmental exposure unit. Ann Allergy Asthma Immunol. 2016 Sep;117(3):310-7. doi: 10.1016/j.anai.2016.07.018. PMID 27613466

RESULTS

PARTICIPANT FLOW:
Groups:
- SPARC Placebo: SPARC Placebo was administered as sprays/nostril QD
- SPARC1310 I: SPARC1310 I was administered as two sprays /nostril QD
- SPARC1310 II: SPARC1310 II was administered as two sprays/nostril QD
- SPARC1310 III: SPARC1310 III was administered as two sprays/nostril QD
Period: Overall Study
Arm/Group | SPARC Placebo | SPARC1310 I | SPARC1310 II | SPARC1310 III
Started | 56 | 55 | 56 | 55
Completed | 55 | 55 | 55 | 53
Not Completed | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- SPARC Placebo; SPARC1310 I: Baseline characteristics: Age
- SPARC1310 II: S0597 mid dose: S0597 mid dose
- SPARC1310 III: S0597 high dose: S0597 high dose
- Total: Total of all reporting groups
Arm/Group | SPARC Placebo | SPARC1310 I | SPARC1310 II | SPARC1310 III | Total
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (10.8) | 39 (9.5) | 39 (10.9) | 38 (10.6) | 39 (10.4)
Age, Customized [Median (Full Range); unit: years] | 38 [18 to 63] | 36 [24 to 59] | 38 [19 to 63] | 37 [19 to 65] | 37 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 29 | 36 | 30 | 136
  Male | 15 | 26 | 20 | 25 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Nasal Symptom Score From Baseline to Day 14.
Description: The 4-point (0=None, 1=Mild, 2=Moderate, and 3=Severe) intensity scale was summed across multiple symptoms (nasal congestion, rhinorrhea, nasal itching, and sneezing). Thus, the TNSS scores could range from 0 to 12, with higher scores indicative of greater severity.
Time Frame: Baseline to Day 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo: Placebo
- S0597 Low Dose: S0597 low dose: S0597 low dose
- S0597 Mid Dose: S0597 mid dose: S0597 mid dose
- S0597 High Dose: S0597 high dose: S0597 high dose
Arm/Group | Placebo | S0597 Low Dose | S0597 Mid Dose | S0597 High Dose
Number analyzed (Participants) | 56 | 55 | 56 | 55
units on a scale | -2.70 (0.381) | -4.05 (0.378) | -4.72 (0.378) | -4.05 (0.385)

ADVERSE EVENTS:
Groups:
- SPARC Placebo: SPARC Placebo administration
- SPARC1310 I: SPARC1310 I administration
- SPARC1310 II: SPARC1310 II administration
- SPARC1310 III: SPARC1310 III administration
Arm/Group | SPARC Placebo | SPARC1310 I | SPARC1310 II | SPARC1310 III
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55 | 0/56 | 0/55
Other Adverse Events (participants affected / at risk) | 2/56 | 3/55 | 4/56 | 4/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPARC Placebo (N=56) | SPARC1310 I (N=55) | SPARC1310 II (N=56) | SPARC1310 III (N=55)
Blood cortisol decreased (Investigations) | 2 | 3 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other